CLINICAL TRIAL: NCT03590860
Title: A Safety, Tolerability, and Pharmacokinetic Study of Single and Multiple Ascending Doses of LY3322207 in Healthy Subjects and Subjects With Hypertension on ACE I/ARB Therapy
Brief Title: A Study of LY3322207 in Healthy Participants and in Participants With Hypertension (High Blood Pressure)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: injection site reaction burden
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16771; I9K-MC-UCAA (Other: Eli Lilly and Company); 2018-002337-38 (EudraCT Number)
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part C will be open label
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY3322207 (Part A) (Experimental): LY3322207 administered subcutaneously (SC)
  Interventions: Drug: LY3322207
- Placebo (Part A) (Placebo Comparator): Placebo matching LY3322207 administered SC
  Interventions: Drug: Placebo
- LY3322207 (Part B) (Experimental): LY3322207 administered SC once weekly
  Interventions: Drug: LY3322207
- Placebo (Part B) (Placebo Comparator): Placebo matching LY3322207 administered SC once weekly
  Interventions: Drug: Placebo
- LY3322207 (Part C) (Experimental): LY3322207 administered SC in participants with hypertension
  Interventions: Drug: LY3322207

INTERVENTIONS:
Drug: LY3322207 — Administered by SC injection
  Arms: LY3322207 (Part A); LY3322207 (Part B); LY3322207 (Part C)
Drug: Placebo — Administered by SC injection
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The purpose of this study is to investigate the safety of the study drug known as LY3322207. Participants must be healthy or must have hypertension (high blood pressure). Participants with hypertension may already be taking a common drug to reduce blood pressure called an angiotensin-converting enzyme inhibitor (ACE-I) or an angiotensin II receptor blocker (ARB).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, as determined by medical history and physical examination, must agree to use a medically appropriate method of birth control and agree not to donate sperm from start of dosing until 90 days beyond last dose
* Healthy females, as determined by medical history and physical examination, of non-child bearing potential due to:

  * Menopause: spontaneous amenorrhea for at least 12 months, not induced by a medical condition such as anorexia nervosa and not taking medications that induced the amenorrhea (for example: oral contraceptives, hormones, gonadotropin releasing hormone, anti-estrogens, selective estrogen receptor modulators, or chemotherapy)
  * Surgical sterilization
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow site specific study procedures
* Have a Body Mass Index (BMI) 18 to 30 kilogram per square meter (kg/m²) at entry
* Have clinical laboratory test results within normal reference range for the population or site, or results with acceptable deviations that are judged not clinically significant
* Be 18 to 55 years old for either Part A or Part B of the study, or 18 to 65 years old for Part C only
* For Part C: must have been treated with a stable dose of ACE-I or ARB for at least 1 month

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 60 days from, a clinical trial involving an investigational drug that has not received regulatory approval
* Have previously completed or withdrawn from this study or any other study investigating this study drug
* Have a history or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, significant atopy, or any clinically significant laboratory abnormality that would preclude study participation
* Have abnormality in the 12-lead electrocardiogram (ECG) which increases study risk
* Have confirmed QT interval corrected by Bazett's method (QTcB) or Fridericia's (QTcF) method >450 millisecond (msec) for men and >470 msec for women
* Have prior Q-wave myocardial infarction or other, specific heart abnormalities, arrhythmias or fibrillations
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure greater than (>)95 or less than (<)50 millimeters of mercury (mmHg) and/or systolic blood pressure >160 or <90 mmHg
* Show evidence of human immunodeficiency virus (HIV), hepatitis C, or hepatitis B
* Have donated blood of more than 100 mL (milliliters) within the last month
* Are unwilling to stop alcohol consumption while resident in the Clinical Research Unit
* Have an average weekly alcohol intake that exceeds 21 units per week (1 unit equal to (=) 12 ounces (oz) or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits)
* Have an abnormal blood pressure (supine) defined as diastolic blood pressure >95 or <50 mmHg and/or systolic blood pressure >160 or <90 mmHg
* Have serum potassium outside normal range
* Have had lymphoma, leukemia, or any malignancy within the past 5 years
* Have clinically significant multiple or severe drug allergies or intolerance
* Are lactating women
* Positive findings for known drugs of abuse
* Have received treatment with biologic agents within 3 months or 5 half-lives prior to dosing
* Participation in any other clinical trial involving a study drug or off-label use of a drug or device, or any other type of medical research judged not to be compatible with this study
* Have estimated glomerular filtration rate (eGFR) < 60 milliliters per minute per 1.73 square meter (mL/min/1.73 m²) for Parts A and B of this study, or eGFR < 50 mL/min/1.73 m² in Part C only
* For Part C: have a history of severe hypertension (defined as SBP greater than or equal to (≥)180 mmHg and/or DBP ≥120 mmHg), secondary hypertension, symptomatic postural hypotension, or hospitalization due to hypertension
* For Part C: have a history of supraventricular tachycardia (for example, atrial fibrillation), ventricular tachycardia, or other cardiac arrhythmia
* For Part C: have resting tachycardia (heart rate ≥100 beats per minute)
* For Part C: have New York Heart Association (NYHA) Class II, III, or IV heart failure, or had any of the following in the previous 3 months: coronary angioplasty, coronary stent placement, coronary bypass surgery or any significant cardiac surgery, myocardial infarction, unstable angina pectoris, cerebrovascular accident, or transient ischemic attack
* For Part C: have an automatic internal cardioverter-defibrillator
* For Part C: have diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Events (Part A) | Baseline up to approximately 31 days
  Serious and other non-serious adverse events will be reported in the Adverse Events Module
Number of Participants with One or More Serious Adverse Events (Part B) | Baseline up to approximately 9 weeks
  Serious and other non-serious adverse events will be reported in the Adverse Events Module
Number of Participants with One or More Serious Adverse Events (Part C) | Baseline up to approximately 9 weeks
  Serious and other non-serious adverse events will be reported in the Adverse Events Module

SECONDARY OUTCOMES:
Area Under the Concentration Versus Time Curve (AUC) of LY3322207 (Part A) | Predose up approximately 31 days
  Pharmacokinetics (PK): AUC of LY3322207
Area Under the Concentration Versus Time Curve (AUC) of LY3322207 (Part B) | Predose up to approximately 9 weeks
  PK: AUC of LY3322207
Area Under the Concentration Versus Time Curve (AUC) of LY3322207 (Part C) | Predose up to approximately 9 weeks
  PK: AUC of LY3322207
Maximum Concentration (Cmax) of LY3322207 (Part A) | Predose up approximately 31 days
  PK: Cmax of LY3322207
Maximum Concentration (Cmax) of LY3322207 (Part B) | Predose up to approximately 9 weeks
  PK: Cmax of LY3322207
Maximum Concentration (Cmax) of LY3322207 (Part C) | Predose up to approximately 9 weeks
  PK: Cmax of LY3322207
Time to reach Cmax (Tmax) of LY3322207 (Part A) | Predose up to approximately Day 31
  PK: Tmax of LY3322207
Time to reach Cmax (Tmax) of LY3322207 (Part B) | Predose up to approximately 9 weeks
  PK: Tmax of LY3322207
Time to reach Cmax (Tmax) of LY3322207 (Part C) | Predose up to approximately 9 weeks
  PK: Tmax of LY3322207
Change from Baseline in Systolic Blood Pressure (SBP) (Part A) | Baseline up approximately 31 days
  Supine position
Change from Baseline in Systolic Blood Pressure (SBP) (Part B) | Baseline up to approximately 9 weeks
  Supine position
Change from Baseline in Systolic Blood Pressure (SBP) (Part C) | Baseline up to approximately 9 weeks
  Supine position
Change from Baseline in Diastolic Blood Pressure (DBP) (Part A) | Baseline up approximately 31 days
  Supine position
Change from Baseline in Diastolic Blood Pressure (DBP) (Part B) | Baseline up to approximately 9 weeks
  Supine position
Change from Baseline in Diastolic Blood Pressure (DBP) (Part C) | Baseline up to approximately 9 weeks
  Supine position
Change from Baseline in Heart Rate (Part A) | Baseline up approximately 31 days
  Supine position
Change from Baseline in Heart Rate (Part B) | Baseline up to approximately 9 weeks
  Supine position
Change from Baseline in Heart Rate (Part C) | Baseline up to approximately 9 weeks
  Supine position

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA Health Sciences, Groningen, Netherlands